CLINICAL TRIAL: NCT06443203
Title: A Randomized Controlled Clinical Trial on Multimodal Prehabilitation in Colorectal Cancer Patients to Improve Functional Capacity and Lower Postoperative Complications.
Brief Title: Multimodal Prehabilitation in Colorectal Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Carlo Feo, Principal Investigator, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 849/2019/Sper/AUSLFe; RF-2018- 12367272 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2024-05-22; First posted 2024-06-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Colon Cancer; Prehabilitation
Keywords: prehabilitation; colorectal surgery; functional capacity; six-minute walking test; post-operative outcomes
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trimodal prehabilitation (Experimental): physical exercise, psychological support and nutritional optimization 4-weeks before surgery
  Interventions: Other: Trimodal prehabilitation
- control group without preoperative prehabilitation (No Intervention): Patients no receiveing prehabilitation and undergoing standard rehabilitation alone after surgery

INTERVENTIONS:
Other: Trimodal prehabilitation — Trimodal prehabilitation program (4-week physical exercise before surgery, nutritional optimization, and psychological support) in patients undergoing ERAS colorectal resection for cancer
  Arms: Trimodal prehabilitation

SUMMARY:
Postoperative complications can occur in up to 50% of individuals undergoing colorectal resection and are associated with poor prognosis, increased costs, and lower health-related quality of life. Even in the absence of complications, after major surgery, patients reduce their physiological and functional capacity by 20-40% and show a higher level of fatigue for 6-8 weeks. Many of these negative effects can be decreased by applying specific ERAS (Enhanced Recovery After Surgery) programs which, by attenuating the neuro-endocrine response induced by surgical trauma, accelerate patients' post-operative convalescence and facilitate their return to functional activities.

In this study, the research group hypothesizes that a prehabilitation program based on physical exercise, nutritional optimization and psychological support (trimodal) carried out by patients in the 4 weeks before elective colorectal resection surgery can determine: 1) better physical performance 8 weeks after surgery (measured by the 6-minute walk test), 2) a possible decrease in postoperative complications, and 3) a reduction in in-hospital (direct) and post-hospital discharge (indirect) costs.

DETAILED DESCRIPTION:
This study aims to determine the effect of prehabilitation on patients' functional capacity and postoperative complications. It is a randomized trial including 112 patients undergoing colorectal surgery for cancer. Patients will be allocated to intervention group receiving 4 weeks trimodal prehabilitation (N=56) or control group receiving no prehabilitation (N=56). After surgery, both groups will follow 8 weeks rehabilitation based on Enhanced Recovery After Surgery (ERAS) guidelines. The primary endpoint is functional capacity, secondary outcomes include postoperative complications and a cost-effectiveness analysis. Multimodal prehabilitation is expected to increase functional capacity and lower postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* patients of age >18 years;
* elective colorectal resection for colonic cancer.

Exclusion Criteria:

* metastatic disease;
* severe walking impairments;
* renal failure stage >2;
* ASA score >3;
* preoperative chemo-radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-06-02 (Estimated); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative functional capacity | From enrollment to the end of treatment at 8 weeks after surgery
  The primary outcome for functional capacity was measured by the 6-Minute Walking Test (6MWT), chosen as a validated, objective measure of colorectal surgery recovery integrating all components of physical activity.

SECONDARY OUTCOMES:
Post-operative complications | Within 30 days after surgery
  To evaluate post-operative complications, the Clavien-Dindo classification has been used as a combined measure of morbidity and mortality.
Hospital length of stay | Within 30 days after surgery
  To evaluate the length of postoperative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Carlo CF Feo, MD FACS, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Unità Operativa Qualità, Accreditamento, Ricerca organizzativa, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bojesen RD, Dalton SO, Skou ST, Jorgensen LB, Walker LR, Eriksen JR, Grube C, Justesen TF, Johansen C, Slooter G, Carli F, Gogenur I. Preoperative multimodal prehabilitation before elective colorectal cancer surgery in patients with WHO performance status I or II: randomized clinical trial. BJS Open. 2023 Nov 1;7(6):zrad134. doi: 10.1093/bjsopen/zrad134. PMID 38060453
- [Background] Molenaar CJL, Minnella EM, Coca-Martinez M, Ten Cate DWG, Regis M, Awasthi R, Martinez-Palli G, Lopez-Baamonde M, Sebio-Garcia R, Feo CV, van Rooijen SJ, Schreinemakers JMJ, Bojesen RD, Gogenur I, van den Heuvel ER, Carli F, Slooter GD; PREHAB Study Group. Effect of Multimodal Prehabilitation on Reducing Postoperative Complications and Enhancing Functional Capacity Following Colorectal Cancer Surgery: The PREHAB Randomized Clinical Trial. JAMA Surg. 2023 Jun 1;158(6):572-581. doi: 10.1001/jamasurg.2023.0198. PMID 36988937
- [Background] Carli F, Charlebois P, Stein B, Feldman L, Zavorsky G, Kim DJ, Scott S, Mayo NE. Randomized clinical trial of prehabilitation in colorectal surgery. Br J Surg. 2010 Aug;97(8):1187-97. doi: 10.1002/bjs.7102. PMID 20602503
- [Background] Gillis C, Fenton TR, Sajobi TT, Minnella EM, Awasthi R, Loiselle SE, Liberman AS, Stein B, Charlebois P, Carli F. Trimodal prehabilitation for colorectal surgery attenuates post-surgical losses in lean body mass: A pooled analysis of randomized controlled trials. Clin Nutr. 2019 Jun;38(3):1053-1060. doi: 10.1016/j.clnu.2018.06.982. Epub 2018 Jul 9. PMID 30025745

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT06443203/Prot_SAP_000.pdf